CLINICAL TRIAL: NCT05147090
Title: Effects of Empagliflozin on Preventing Fibrosis and Cirrhosis Progression in Nucleos(t)Ide Analogue-treated Chronic Hepatitis B Patients With F2-F4 Fibrosis: a Randomized, Double-blind Placebo-controlled Trial
Brief Title: Effects of Empagliflozin on Fibrosis and Cirrhosis in Chronic Hepatitis B Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Research Grant Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW-21023
Record Dates: First submitted 2021-11-22; First posted 2021-12-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis b; NAFLD; Cirrhosis; Fibrosis, Liver; Empagliflozin; SGLT2 Inhibitors
MeSH Terms: conditions — Hepatitis B, Chronic; Non-alcoholic Fatty Liver Disease; Fibrosis; Liver Cirrhosis | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomly allocated to either the empagliflozin group or placebo group (i.e. control group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo pills will be manufactured in identical appearance to the study drug (empagliflozin)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin group (Active Comparator): Empagliflozin 10mg daily for 156 weeks
  Interventions: Drug: Empagliflozin 10 MG
- Placebo group (Placebo Comparator): Placebo pills (identical in appearance to empagliflozin 10mg) daily for 156 weeks
  Interventions: Drug: Placebo pills

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Empagliflozin 10mg daily
  Other Names: empagliflozin
  Arms: Empagliflozin group
Drug: Placebo pills — Identical in appearance to empagliflozin 10mg daily
  Other Names: placebo
  Arms: Placebo group

SUMMARY:
Chronic hepatitis B (CHB) affects 257million individuals worldwide. In 2017, it caused around 39.7 million cases of cirrhosis and 0.4 million cirrhosis-related deaths in 2017. However, there is no specific treatment for liver fibrosis/cirrhosis. Although nucleos(t)ide analogues (NAs) profoundly suppress viral replication, fibrosis/cirrhosis progression can still occur in NA-treated patients.

Sodium-glucose cotransporter type-2 (SGLT2) inhibitors are antidiabetic drugs that may prevent fibrosis/cirrhosis progression by reducing hepatic steatosis/inflammation, dampening renin-angiotensin aldosterone system (RAAS) activation, and reducing fluid retention, effects of which are independent of glycemic control. Clinical studies in diabetic patients show SGLT2 inhibitors reduce hepatis steatosis/inflammation, regress ascites (a cirrhotic complication), and improve liver function parameters and survival prognosis in terms of model for end-stage liver disease (MELD) score. There are currently no randomized controlled trials (RCTs) on role of SGLT2 inhibitors in preventing fibrosis/cirrhosis progression in CHB patients. Magnetic resonance elastography (MRE) and transient elastography (TE) are non-invasive techniques for liver stiffness measurement (LSM), although MRE is more accurate than TE.

The investigators propose a double-blind, randomized, placebo-controlled trial to compare effect of empagliflozin (an SGLT2 inhibitor) with placebo (1:1 ratio) in preventing fibrosis progression in both diabetic and non-diabetic NA-treated CHB patients with significant/advanced fibrosis or compensated cirrhosis. 108 patients will be randomly sampled from our pre-existing TE database. Empagliflozin 10mg daily will be given to treatment arm. Placebo pills will be manufactured identical in appearance to empagliflozin. Subjects will receive active or placebo pills for three years, and undergo clinical, anthropometric and laboratory assessments (at baseline, weeks 8, 16, and every 4 months thereafter). They will undergo LSM by TE at baseline, end of first, second and third year, and by MRE at baseline and end of third year. Primary outcome is difference in change to liver stiffness (measured by MRE) from baseline between the two groups at the end of third year.

The study results will determine whether SGLT2 inhibitors can prevent hepatic fibrosis/cirrhosis progression in NA-treated CHB patients.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) affects 257million individuals worldwide. In 2017, it caused around 39.7 million cases of cirrhosis and 0.4 million cirrhosis-related deaths in 2017. However, there is no specific treatment for liver fibrosis/cirrhosis. Although nucleos(t)ide analogues (NAs) profoundly suppress viral replication, fibrosis/cirrhosis progression can still occur in NA-treated patients.

Sodium-glucose cotransporter type-2 (SGLT2) inhibitors are antidiabetic drugs that may prevent fibrosis/cirrhosis progression by reducing hepatic steatosis/inflammation, dampening renin-angiotensin aldosterone system (RAAS) activation, and reducing fluid retention, effects of which are independent of glycemic control. Clinical studies in diabetic patients show SGLT2 inhibitors reduce hepatis steatosis/inflammation, regress ascites (a cirrhotic complication), and improve liver function parameters and survival prognosis in terms of model for end-stage liver disease (MELD) score. Our preliminary data from a territory-wide electronic healthcare database shows SGLT2 inhibitors were associated with 58% reduction in risk of cirrhosis development over three years among CHB patients with diabetes (n=9,502). There are currently no randomized controlled trials (RCTs) on role of SGLT2 inhibitors in preventing fibrosis/cirrhosis progression in CHB patients. Magnetic resonance elastography (MRE) and transient elastography (TE) are non-invasive techniques for liver stiffness measurement (LSM), although MRE is more accurate than TE.

The novelty of utilizing "drug repositioning" by changing role of SGLT2 inhibitors in treating diabetes mellitus (DM) to preventing fibrosis/cirrhosis progression in CHB deserves exploration. We propose a double-blind, randomized, placebo-controlled trial to compare effect of empagliflozin (an SLGT2 inhibitor) with placebo (1:1 ratio) in reducing liver stiffness in both diabetic and non-diabetic NA-treated CHB patients with significant/advanced fibrosis or compensated cirrhosis. 108 patients will be randomly sampled from our pre-existing TE database. Empagliflozin 10mg daily will be given to treatment arm. Placebo pills will be manufactured identical in appearance to empagliflozin. Subjects will receive active or placebo pills for three years, and undergo clinical, anthropometric and laboratory assessments (at baseline, weeks 8, 16, and every 4 months thereafter). They will undergo LSM by TE at baseline, end of first, second and third year, and by MRE at baseline and end of third year. Primary outcome is difference in change to liver stiffness (measured by MRE) from baseline between the two groups at the end of third year. Secondary outcomes are remission of advanced fibrosis/cirrhosis, progression of advanced fibrosis to cirrhosis, improvement of laboratory results (liver transaminases, ferritin, glucose, lipid profiles) and anthropometric measurements.

The study results will determine whether SGLT2 inhibitors can prevent hepatic fibrosis/cirrhosis progression in NA-treated CHB patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited if they have significant/advanced fibrosis or cirrhosis confirmed by MRE

Exclusion Criteria:

1. decompensated cirrhosis (variceal bleeding, ascites, hepatic hydrothorax, hepatic encephalopathy),
2. portal vein thrombosis,
3. alcohol intake >20g within last 2 years,
4. concurrent chronic liver disease (chronic hepatitis C infection, autoimmune hepatitis, Wilson's disease, hemochromatosis, primary biliary cholangitis, drug-induced),
5. history of malignancy including hepatocellular carcinoma (HCC),
6. pregnancy,
7. contraindications to empagliflozin (estimated glomerular filtration rate (eGFR) <45mL/min/1.73m2, recurrent genitourinary tract infections, gangrene, allergy),
8. contraindications to MRI (e.g., claustrophobia, implanted devices with ferromagnetic properties).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in liver stiffness (measured by MRE) | week 156
  difference in change to liver stiffness from baseline between the two groups at the end of year 3 as measured by MRE

SECONDARY OUTCOMES:
Remission of significant/advanced fibrosis and cirrhosis | week 156
  Remission of advanced fibrosis and cirrhosis (defined as a decrease in 1 fibrosis stage using MRE) at the end of year 3
Progression of significant/advanced fibrosis to cirrhosis (measured by MRE) | week 156
  Progression of significant/advanced fibrosis to cirrhosis (as defined by MRE) at the end of year 3
Progression to decompensated cirrhosis | week 156
  Progression to decompensated cirrhosis (ascites, variceal bleeding and/or hepatic encephalopathy) at the end of year 3
Change in liver stiffness (measured by transient elastography) | week 26, 52, 104 and 156
  Difference in serial changes to liver stiffness from baseline between the two groups (LSM measured by transient elastography)
Change in fat content (measured by transient elastography) | week 26, 52, 104 and 156
  Difference in serial changes to liver fat content from baseline between the two groups (CAP measured by transient elastography)
Changes of alanine aminotransferase (ALT) | week 26, 52, 104 and 156
  Changes of ALT at week 26, 52, 104 and 156
Changes of aspartate aminotransferase (AST) | week 26, 52, 104 and 156
  Changes of AST at week 26, 52, 104 and 156
Changes of alkaline phosphatase (ALP) | week 26, 52, 104 and 156
  Changes of ALP at week 26, 52, 104 and 156
Changes of gamma glutamyl transferase (GGT) | week 26, 52, 104 and 156
  Changes of GGT at week 26, 52, 104 and 156
Changes of fasting glucose | week 26, 52, 104 and 156
  Changes of fasting glucose at week 26, 52, 104 and 156
Changes of haemoglobin A1c (HbA1c) | week 26, 52, 104 and 156
  Changes of HbA1c at week 26, 52, 104 and 156
Changes of total cholesterol | week 26, 52, 104 and 156
  Changes of total cholesterol at week 26, 52, 104 and 156
Changes of low density lipoprotein (LDL) | week 26, 52, 104 and 156
  Changes of LDL at week 26, 52, 104 and 156
Changes of high density lipoprotein (HDL) | week 26, 52, 104 and 156
  Changes of HDL at week 26, 52, 104 and 156
Changes of body weight | week 26, 52, 104 and 156
  Changes of body weight at week 26, 52, 104 and 156
Changes of body mass index (BMI) | week 26, 52, 104 and 156
  Changes of BMI at week 26, 52, 104 and 156
Changes of waist circumference | week 26, 52, 104 and 156
  Changes of waist circumference at week 26, 52, 104 and 156
Changes of systolic blood pressure | week 26, 52, 104 and 156
  Changes of systolic blood pressure at week 26, 52, 104 and 156
Changes of diastolic blood pressure | week 26, 52, 104 and 156
  Changes of diastolic blood pressure at week 26, 52, 104 and 156

CONTACTS AND LOCATIONS:
Overall Officials: Ka Shing Cheung, MD, MPH, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong/Queen Mary Hospital, Hong Kong, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be made available in the form of excel files upon request by other researchers